CLINICAL TRIAL: NCT06756061
Title: A Nation-wide, Multi-center, Prospective, Randomized, Parallel-group, Open-label, Investigator Initiated Pilot Study to Evaluate Efficacy and Safety of Systemic Corticosteroid Plus Ruxolitinib as First-line Therapy in Patients With New-onset Moderate to Severe Chronic Graft-versus-host Disease
Brief Title: Comparing the Therapeutic Effects of Using Ruxolitinib and Steroids Concurrently to Steroids Alone as Initial Treatment In Patients Diagnosed With Chronic Graft-versus-host Disease at a Grade of Moderate or Higher Severity
Acronym: FRONTJAK-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Byung-Sik Cho (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Byung-Sik Cho, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424DKR01T
Record Dates: First submitted 2024-12-13; First posted 2025-01-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: GVHD - Graft-Versus-Host Disease; Neoplasms; Haematopoietic Stem Cell Transplantation
Keywords: GvHD-Graft-Versus-Host-Disease; ruxolitinib; first-line
MeSH Terms: conditions — Graft vs Host Disease; Neoplasms | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone + Jakavi(ruxolitinib) (Experimental): The experimental group will receive ruxolitinib 10 mg orally twice daily (BID) and prednisone (or equivalent) at a dosage of 1 mg/kg/day.
  Subjects are orally administered with an investigational medicinal product (IMP) according to their designated treatment group for 48 weeks, and the investigator may adjust the dosage of IMPs based on symptoms of the target disease. (However, after the 48-week mark, participants in the ruxolitinib treatment group may continue to receive ruxolitinib for an additional maximum of 2 years, based on the investigator's judgment regarding the need for ongoing treatment. The total duration of ruxolitinib administration will not exceed 3 years.)
  Interventions: Drug: Prednisone + Jakavi(ruxolitinib)
- Prednisone (Active Comparator): The control group will receive prednisone (or equivalent) at a dosage of 1 mg/kg/day.
  Subjects are orally administered with an investigational medicinal product (IMP) according to their designated treatment group for 48 weeks, and the investigator may adjust the dosage of IMPs based on symptoms of the target disease.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone + Jakavi(ruxolitinib) — The experimental group will receive ruxolitinib 10 mg orally twice daily (BID) and prednisone (or equivalent) at a dosage of 1 mg/kg/day.
  Subjects are orally administered with an investigational medicinal product (IMP) according to their designated treatment group for 48 weeks, and the investigator may adjust the dosage of IMPs based on symptoms of the target disease. (However, after the 48-week mark, participants in the ruxolitinib treatment group may continue to receive ruxolitinib for an additional maximum of 2 years, based on the investigator's judgment regarding the need for ongoing treatment. The total duration of ruxolitinib administration will not exceed 3 years.)
  Arms: Prednisone + Jakavi(ruxolitinib)
Drug: Prednisone — The control group will receive prednisone (or equivalent) at a dosage of 1 mg/kg/day.
  Subjects are orally administered with an investigational medicinal product (IMP) according to their designated treatment group for 48 weeks, and the investigator may adjust the dosage of IMPs based on symptoms of the target disease.
  Arms: Prednisone

SUMMARY:
Chronic graft-versus-host disease (cGVHD) is a complication that occurs in 30-40% of recipients of allogeneic hematopoietic stem cell transplantation (allo-HSCT) and is a major cause of late non-relapse mortality. In cases where the initial treatment response is inadequate, irreversible tissue damage often persists, making it a fatal complication that significantly reduces quality of life even for long-term survivors.

Therefore, the success of first-line treatment is crucial, but to date, there are no approved drugs specifically for the first-line treatment of chronic graft-versus-host disease. Besides corticosteroids, which have been used palliatively for over 50 years, there are no proven effective treatments available.

Against this background, this study was designed to explore the potential of new treatments as first-line therapy for chronic graft-versus-host disease, where effective treatment options are currently lacking.

Initially, the objective response rate will be analyzed at the 48-week mark based on the NIH Consensus Criteria (Lee 2015). Additionally, the study will evaluate the proportion of patients with steroid-resistant or steroid-dependent conditions, the objective response rate(ORR), failure-free survival(FFS), duration of response(DOR), and the proportion of patients who have reduced corticosteroids. Furthermore, the differences in treatment effects between the two groups of patients will be analyzed based on safety endpoints, including adverse events, laboratory tests, physical examinations, and vital signs.

ELIGIBILITY:
[Inclusion Data]

1. Adult men and women aged 19 or older based on the date of signing on the informed consent form
2. On the screening visit, those who are diagnosed of a moderate to severe chronic graft-versus-host disease according to 2014 NIH consensus criteria

   -Moderate: At least one of the following conditions: >1 point for at least three organs >2 points for at least one organ except the lungs >1 point for the lungs

   -Severe: At least one of the following conditions: >3 points for at least one organ
   * At least 2 points for the lungs
3. Those who have no history of systemic treatment for chronic graft-versus-host disease and now need systemic corticosteroid treatment
4. Those whose ECOG (Eastern Cooperative Oncology Group) performance status is 0 to 2.
5. Regardless of the donor (matched sibling-family donor, matched unrelated donor, or partially matched family donor), those who have successfully taken same-type stem cell transplantation (alloSCT) from the marrow, peripheral blood stem cell, or cord blood
6. Those who voluntarily agree on participation in this clinical trial

[Exclusion Data]

1. Those who meet the following criteria in laboratory tests during the screening and randomization visits

   * Those whose platelet count is less than or equal to 25,000/mm3 without blood transfusion
   * Those whose absolute neutrophil count is less than or equal to 1,000/mm3
   * Those whose total bilirubin > 3 x ULN for any reason other than chronic graft-versus-host disease
2. Those with gastrointestinal troubles that hinder the intake and absorption of IMPs and concomitant medicines (systemic corticosteroid) (e.g.: signs such as ulcerative disease, unregulated nausea, vomiting, diarrhea, malabsorption, etc. or small intestine removal)
3. Those with a history of graft-versus-host disease treatment

   * Corticosteroid administration is permitted for chronic graft-versus-host disease treatment within 72 hours before the randomization visit
   * Except those who had therapeutic or preventive use of systemic corticosteroids and/or systemic immunosuppressants (CNI, MMF) for acute graft-versus-host disease (In case of prednisone administration for maintenance, only 0.5 mg/kg/day or less is permitted)
4. Those to whom the treatment for chronic graft-versus-host disease cannot begin as prednisone ≥ 0.5 mg/kg/day
5. Those whose same-type stem cell transplantation (alloSCT) has been confirmed as engraft-failed within 6 months before the screening visit
6. Those with an experience of ruxolitinib administration for acute graft-versus-host disease treatment (however, the patient may participate on the assumption that the response to the acute graft-versus-host disease treatment reaches the level of complete or partial response and that there is no ruxolitinib administration history within 4 weeks before the randomization visit. In addition, if ruxolitinib administration was for another disease, the patient may participate unless there is no history of ruxolitinib administration within 4 weeks before the randomization visit.)
7. Those who suffer chronic graft-versus-host disease after an unscheduled donor lymphocyte infusion for proactive treatment to prevent the recurrence of a malignant tumor (Participation is allowed if the scheduled lymphocyte infusion is performed as part of the transplantation procedure, not for the prevention of the recurrence of a malignant tumor.)
8. Those found to have the following history in the screening visit:

   * Relapsed primary malignancy
   * Those found to involve an unregulated sinusoidal obstruction syndrome
   * Those with a history of progressive multifocal leukoencephalopathy (PML)
   * Nephropathy whose creatinine clearance rate is lower than 30 mL/min (Cockroft Gault equation)
   * Infections that are clinically active and uncontrolled, requiring treatment, including significant bacteria, fungi, viruses, or parasitic infections. (However, if there are no signs of progression at the time of screening due to appropriate treatment, the infection is considered controlled. The progression of infection is defined by hemodynamic instability due to sepsis, new symptoms caused by the infection, worsening physical signs, or radiological findings. A persistent fever without other signs or symptoms is not interpreted as progressive infection.)
   * Active tuberculosis
   * HIV-infected individual
   * Active infection of hepatitis B virus (HBV) or hepatitis C virus (HCV) that the investigator views as significant
   * Cardiovascular disease that the investigator considers as clinically significant (acute cardiac infarction (within 6 months before randomization), NYHA class III or IV congestive heart failure, unstable angina (within 6 months before randomization), clinically significant symptomatic cardiac arrhythmia (e.g.: continued ventricular tachycardia, clinically significant level 2 or 3 AV blockage with no pacemaker used), unregulated hypertension)
9. Those allergic or sensitive to additives of IMPs and concomitant medicines (systemic corticosteroid) or similar compounds
10. Patients with genetic problems such as galactose intolerance, lapp lactase deficiency, glucose - galactose malabsorption, etc.
11. Those who are administrated with more than 200 mg of Fluconazole per day
12. Those being treated with systemic medicines that may hinder blood coagulation or platelet functions such as aspirin, heparin, and warfarin (However, those whose aspirin administration does not exceed 150 mg/day may participate.)
13. Pregnant or breast-feeding women
14. Those who do not agree on utilizing proper methods of contraception(e.g. a copper intrauterine device (copper loop), an intrauterine device containing hormones, condoms, a vasectomy, tubal surgery, a spermicide, a vagina-inserted contraceptive, a subdermal implant, an injectable contraceptive, a female condom, oral contraceptive, etc.) during the period of this clinical trial(the period of IP administration and at least 30 days after IP administration ends)
15. Those who have participated in another clinical trial within 30 days before the screening visit and have a history of IMP administration/medical equipment application (However, if the investigator views such a previous trial as not affecting this clinical trial's efficacy and safety assessment such as observational study or retrospective study, the subject may participate.)
16. Those whose participation in this clinical trial is viewed as inappropriate in the investigator's opinion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | on 48 week
  ORR was defined as the proportion of participants in each study arm achieving either a complete response (CR) or partial response (PR) based on chronic GvHD (cGvHD) assessments in accordance with the National Institutes of Health Consensus Criteria. Response scoring was compared against the organ score at the time of randomization. CR was characterized by the complete resolution of all cGvHD-related signs and symptoms across all evaluable organs, without the initiation or addition of new systemic therapies. PR was defined as improvement in at least one organ (e.g., an increase of 1 or more points on a 4- to 7-point scale, or an increase of 2 or more points on a 10- to 12-point scale) with no progression in other organs or sites and without the need for initiation or addition of new systemic therapies. Participants requiring additional systemic therapies for earlier progression, mixed response, or non-response were classified as not achieving response.

SECONDARY OUTCOMES:
Ratio of subjects who are found steroid-refractory or steroid-dependent | on Weeks 1, 4, 24, 36 and 48
  All corticosteroid dosages administered to participants, along with any dose adjustments made during the study, were documented to evaluate participants meeting specific criteria.Steroid-refractory chronic GvHD(SR-cGVHD) was defined as either progression of cGVHD while receiving prednisone at a dose of ≥1mg/kg/day for at least 1 week or stable cGVHD while on≥0.5mg/kg/day or ≥1mg/kg every other day(EOD) for at least 1 month.Response criteria were based on the National Institutes of Health Consensus Criteria.Progression was defined as worsening in any organ or site or the need to initiate or add new systemic therapies.Participants who did not meet the criteria for overall response or progression were categorized as stable.Steroid-dependent participants were defined as those for whom at least two corticosteroid tapering attempts, spaced at least 8 weeks apart, had failed, requiring corticosteroid doses>0.25 mg/kg/day or >0.5mg/kg/day EOD to prevent recurrence or progression of symptoms.
Overall Response Rate (ORR) based on the NIH Consensus Criteria on Weeks 24 and 36 | on Weeks 24 and 36
  ORR was defined as the proportion of participants in each study arm achieving either a complete response (CR) or partial response (PR) based on chronic GvHD (cGvHD) assessments in accordance with the National Institutes of Health Consensus Criteria. Response scoring was compared against the organ score at the time of randomization. CR was characterized by the complete resolution of all cGvHD-related signs and symptoms across all evaluable organs, without the initiation or addition of new systemic therapies. PR was defined as improvement in at least one organ (e.g., an increase of 1 or more points on a 4- to 7-point scale, or an increase of 2 or more points on a 10- to 12-point scale) with no progression in other organs or sites and without the need for initiation or addition of new systemic therapies. Participants requiring additional systemic therapies for earlier progression, mixed response, or non-response were classified as not achieving response.
Failure-free Survival (FFS) | for 48 weeks
  Composite time to event endpoint incorporating the following FFS events: (i) relapse or recurrence of underlying disease or death due to underlying disease, (ii) nonrelapse mortality, or (iii) addition or initiation of another systemic therapy for cGvHD.
Duration of Response (DOR) | for 48 weeks
  DOR was defined as the time from first response until cGvHD progression, death, or the date of change/addition of systemic therapies for cGvHD and as assessed for responders only. Response was based on cGvHD disease assessments (National Institutes of Health consensus criteria). Duration of response was evaluated in participants who achieved a CR or PR at or before Cycle 7 Day 1.
Ratio of subjects whose daily dosage of systemic corticosteroid is reduced as much as at least 50% | compared to the baseline on Week 48
  All corticosteroid dosages administered to participants, along with any dose adjustments made during the study, were documented to evaluate participants who achieved a ≥ 50% reduction in their daily corticosteroid dose.
Ratio of subjects whose daily dosage of systemic corticosteroid is reduced | compared to the baseline on Week 48
  All corticosteroid dosages administered to participants, along with any dose adjustments made during the study, were documented for assessment of participants with any degree of reduction in daily corticosteroid dose.
Time up to the point of stopping systemic immunosuppressant administration (concomitant medicines other than IMPs) | for 48 weeks
  All systemic immunosuppressant dosages administered to participants, along with any dose adjustments during the study, were documented to assess participants who successfully discontinued all systemic immunosuppressants. Participants who were classified as having completely tapered off immunosuppressants were those who permanently ceased their use as recorded in the dose administration records and did not restart treatment within the same interval. Participants who discontinued immunosuppressants and remained in follow-up were also considered tapered off, with a recorded dose of 0 in subsequent intervals unless they restarted immunosuppressant treatment or withdrew from the main treatment period.
Change in FACT-BMT((Functional Assessment of Cancer Therapy - Bone Marrow Transplantation) score | compared to the baseline on Week 24, 36 and 48
  Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The FACT-BMT is a 50-item self-report questionnaire that measures the effect of a therapy on domains including physical, functional, social/family, and emotional well-being, together with additional concerns relevant for bone marrow transplantation participants. The questions were based on a 5-point Likert scale, where 0 corresponds to "not at all" and 4 corresponds to "very much." The higher the final score, the better the quality of life. The FACT-BMT total score ranges from 0 to 148.
Change in EQ-5D-5L(European Quality of Life 5 Dimension) score | compared to the baseline on Week 24, 36 and 48
  The EQ-5D-5L is a descriptive classification consisting of five dimensions of health: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. The five-level version (no problems, slight problems, moderate problems, severe problems, and extreme problems) uses a 5-point Likert scale, with 1 being no problems and 5 being extreme problems.

OTHER OUTCOMES:
Number of Participants With Any Treatment-emergent Adverse Event (TEAE) | for 48 weeks
  Adverse events (AEs) were defined as the onset or worsening of any undesirable signs, symptoms, or medical conditions that occurred after the participant provided signed informed consent. Abnormal laboratory values or test results following informed consent were classified as AEs only if they resulted in clinical signs or symptoms, were deemed clinically significant, required intervention (e.g., treatment for hematologic abnormalities such as transfusion or hematopoietic stem cell support), or necessitated changes in study medication(s). Treatment-emergent adverse events (TEAEs) were defined as AEs that began or worsened during the on-treatment period, which included both the randomized and cross-over phases of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Banpo-daero/Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeFilipp Z, Couriel DR, Lazaryan A, Bhatt VR, Buxbaum NP, Alousi AM, Olivieri A, Pulanic D, Halter JP, Henderson LA, Zeiser R, Gooley TA, MacDonald KPA, Wolff D, Schultz KR, Paczesny S, Inamoto Y, Cutler CS, Kitko CL, Pidala JA, Lee SJ, Socie G, Sarantopoulos S, Pavletic SZ, Martin PJ, Blazar BR, Greinix HT. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: III. The 2020 Treatment of Chronic GVHD Report. Transplant Cell Ther. 2021 Sep;27(9):729-737. doi: 10.1016/j.jtct.2021.05.004. Epub 2021 Jun 11. PMID 34147469
- [Background] Martin PJ, Lee SJ, Przepiorka D, Horowitz MM, Koreth J, Vogelsang GB, Walker I, Carpenter PA, Griffith LM, Akpek G, Mohty M, Wolff D, Pavletic SZ, Cutler CS. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. The 2014 Clinical Trial Design Working Group Report. Biol Blood Marrow Transplant. 2015 Aug;21(8):1343-59. doi: 10.1016/j.bbmt.2015.05.004. Epub 2015 May 15. PMID 25985921
- [Background] Malard F, Labopin M, Yakoub-Agha I, Chantepie S, Guillaume T, Blaise D, Tabrizi R, Magro L, Vanhove B, Blancho G, Moreau P, Gaugler B, Chevallier P, Mohty M. Rituximab-based first-line treatment of cGVHD after allogeneic SCT: results of a phase 2 study. Blood. 2017 Nov 16;130(20):2186-2195. doi: 10.1182/blood-2017-05-786137. Epub 2017 Sep 1. PMID 28864814
- [Background] Rongvaux-Gaida D, Dupuis M, Poupon J, Djebrani-Oussedik N, Lemonnier C, Rieger F. High Response Rate and Corticosteroid Sparing with Arsenic Trioxide-Based First-Line Therapy in Chronic Graft-versus-Host Disease after Allogeneic Hematopoietic Stem Cell Transplantation. Transplant Cell Ther. 2022 Oct;28(10):679.e1-679.e11. doi: 10.1016/j.jtct.2022.07.004. Epub 2022 Jul 10. PMID 35830931
- [Background] Lazaryan A, Lee S, Arora M, Kim J, Betts BC, Khimani F, Nishihori T, Bejanyan N, Liu H, Kharfan-Dabaja MA, Locke FL, Gonzalez R, Jain MD, Davila ML, Perez LE, Mishra A, Perez Perez A, Balke K, Ayala E, Ochoa L, Castaneda Puglianini O, Faramand R, Alsina M, Elmariah H, Nieder ML, Fernandez H, Anasetti C, Pidala JA. A phase 2 multicenter trial of ofatumumab and prednisone as initial therapy for chronic graft-versus-host disease. Blood Adv. 2022 Jan 11;6(1):259-269. doi: 10.1182/bloodadvances.2021005552. PMID 34649279
- [Background] Zeiser R, von Bubnoff N, Butler J, Mohty M, Niederwieser D, Or R, Szer J, Wagner EM, Zuckerman T, Mahuzier B, Xu J, Wilke C, Gandhi KK, Socie G; REACH2 Trial Group. Ruxolitinib for Glucocorticoid-Refractory Acute Graft-versus-Host Disease. N Engl J Med. 2020 May 7;382(19):1800-1810. doi: 10.1056/NEJMoa1917635. Epub 2020 Apr 22. PMID 32320566
- [Background] Martin PJ, Storer BE, Rowley SD, Flowers ME, Lee SJ, Carpenter PA, Wingard JR, Shaughnessy PJ, DeVetten MP, Jagasia M, Fay JW, van Besien K, Gupta V, Kitko C, Johnston LJ, Maziarz RT, Arora M, Jacobson PA, Weisdorf D. Evaluation of mycophenolate mofetil for initial treatment of chronic graft-versus-host disease. Blood. 2009 May 21;113(21):5074-82. doi: 10.1182/blood-2009-02-202937. Epub 2009 Mar 6. PMID 19270260
- [Background] Hamilton BK. Updates in chronic graft-versus-host disease. Hematology Am Soc Hematol Educ Program. 2021 Dec 10;2021(1):648-654. doi: 10.1182/hematology.2021000301. PMID 34889364
- [Background] Lee SJ, Vogelsang G, Flowers ME. Chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2003 Apr;9(4):215-33. doi: 10.1053/bbmt.2003.50026. PMID 12720215
- [Background] Flowers ME, Martin PJ. How we treat chronic graft-versus-host disease. Blood. 2015 Jan 22;125(4):606-15. doi: 10.1182/blood-2014-08-551994. Epub 2014 Nov 14. PMID 25398933
- [Background] Axt L, Naumann A, Toennies J, Haen SP, Vogel W, Schneidawind D, Wirths S, Moehle R, Faul C, Kanz L, Axt S, Bethge WA. Retrospective single center analysis of outcome, risk factors and therapy in steroid refractory graft-versus-host disease after allogeneic hematopoietic cell transplantation. Bone Marrow Transplant. 2019 Nov;54(11):1805-1814. doi: 10.1038/s41409-019-0544-y. Epub 2019 May 14. PMID 31089279
- [Background] Koc S, Leisenring W, Flowers ME, Anasetti C, Deeg HJ, Nash RA, Sanders JE, Witherspoon RP, Storb R, Appelbaum FR, Martin PJ. Therapy for chronic graft-versus-host disease: a randomized trial comparing cyclosporine plus prednisone versus prednisone alone. Blood. 2002 Jul 1;100(1):48-51. doi: 10.1182/blood.v100.1.48. PMID 12070007
- [Background] Arora M, Wagner JE, Davies SM, Blazar BR, Defor T, Enright H, Miller WJ, Weisdorf DF. Randomized clinical trial of thalidomide, cyclosporine, and prednisone versus cyclosporine and prednisone as initial therapy for chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2001;7(5):265-73. doi: 10.1053/bbmt.2001.v7.pm11400948.
- [Background] Penack O, Marchetti M, Ruutu T, Aljurf M, Bacigalupo A, Bonifazi F, Ciceri F, Cornelissen J, Malladi R, Duarte RF, Giebel S, Greinix H, Holler E, Lawitschka A, Mielke S, Mohty M, Arat M, Nagler A, Passweg J, Schoemans H, Socie G, Solano C, Vrhovac R, Zeiser R, Kroger N, Basak GW. Prophylaxis and management of graft versus host disease after stem-cell transplantation for haematological malignancies: updated consensus recommendations of the European Society for Blood and Marrow Transplantation. Lancet Haematol. 2020 Feb;7(2):e157-e167. doi: 10.1016/S2352-3026(19)30256-X. PMID 32004485
- [Background] Pidala J, Kurland B, Chai X, Majhail N, Weisdorf DJ, Pavletic S, Cutler C, Jacobsohn D, Palmer J, Arai S, Jagasia M, Lee SJ. Patient-reported quality of life is associated with severity of chronic graft-versus-host disease as measured by NIH criteria: report on baseline data from the Chronic GVHD Consortium. Blood. 2011 Apr 28;117(17):4651-7. doi: 10.1182/blood-2010-11-319509. Epub 2011 Feb 25. PMID 21355084
- [Background] DeFilipp Z, Alousi AM, Pidala JA, Carpenter PA, Onstad LE, Arai S, Arora M, Cutler CS, Flowers MED, Kitko CL, Chen GL, Lee SJ, Hamilton BK. Nonrelapse mortality among patients diagnosed with chronic GVHD: an updated analysis from the Chronic GVHD Consortium. Blood Adv. 2021 Oct 26;5(20):4278-4284. doi: 10.1182/bloodadvances.2021004941. PMID 34521116
- [Background] Cho BS, Lee SE, Song HH, Lee JH, Yahng SA, Eom KS, Kim YJ, Kim HJ, Lee S, Min CK, Cho SG, Kim DW, Lee JW, Min WS, Park CW. Graft-versus-tumor effect according to type of graft-versus-host disease defined by National Institutes of Health consensus criteria and associated outcomes. Biol Blood Marrow Transplant. 2012 Jul;18(7):1136-43. doi: 10.1016/j.bbmt.2012.01.010. Epub 2012 Jan 16. PMID 22261380
- [Background] Kondo M, Kojima S, Horibe K, Kato K, Matsuyama T. Risk factors for chronic graft-versus-host disease after allogeneic stem cell transplantation in children. Bone Marrow Transplant. 2001 Apr;27(7):727-30. doi: 10.1038/sj.bmt.1702868. PMID 11360113
- [Background] Arai S, Arora M, Wang T, Spellman SR, He W, Couriel DR, Urbano-Ispizua A, Cutler CS, Bacigalupo AA, Battiwalla M, Flowers ME, Juckett MB, Lee SJ, Loren AW, Klumpp TR, Prockup SE, Ringden OT, Savani BN, Socie G, Schultz KR, Spitzer T, Teshima T, Bredeson CN, Jacobsohn DA, Hayashi RJ, Drobyski WR, Frangoul HA, Akpek G, Ho VT, Lewis VA, Gale RP, Koreth J, Chao NJ, Aljurf MD, Cooper BW, Laughlin MJ, Hsu JW, Hematti P, Verdonck LF, Solh MM, Norkin M, Reddy V, Martino R, Gadalla S, Goldberg JD, McCarthy PL, Perez-Simon JA, Khera N, Lewis ID, Atsuta Y, Olsson RF, Saber W, Waller EK, Blaise D, Pidala JA, Martin PJ, Satwani P, Bornhauser M, Inamoto Y, Weisdorf DJ, Horowitz MM, Pavletic SZ; Graft-vs-Host Disease Working Committee of the CIBMTR. Increasing incidence of chronic graft-versus-host disease in allogeneic transplantation: a report from the Center for International Blood and Marrow Transplant Research. Biol Blood Marrow Transplant. 2015 Feb;21(2):266-74. doi: 10.1016/j.bbmt.2014.10.021. Epub 2014 Oct 30. PMID 25445023
- [Background] Zeiser R, Blazar BR. Pathophysiology of Chronic Graft-versus-Host Disease and Therapeutic Targets. N Engl J Med. 2017 Dec 28;377(26):2565-2579. doi: 10.1056/NEJMra1703472. No abstract available. PMID 29281578
- [Background] Jagasia MH, Greinix HT, Arora M, Williams KM, Wolff D, Cowen EW, Palmer J, Weisdorf D, Treister NS, Cheng GS, Kerr H, Stratton P, Duarte RF, McDonald GB, Inamoto Y, Vigorito A, Arai S, Datiles MB, Jacobsohn D, Heller T, Kitko CL, Mitchell SA, Martin PJ, Shulman H, Wu RS, Cutler CS, Vogelsang GB, Lee SJ, Pavletic SZ, Flowers ME. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015 Mar;21(3):389-401.e1. doi: 10.1016/j.bbmt.2014.12.001. Epub 2014 Dec 18. PMID 25529383
- [Background] Spoerl S, Mathew NR, Bscheider M, Schmitt-Graeff A, Chen S, Mueller T, Verbeek M, Fischer J, Otten V, Schmickl M, Maas-Bauer K, Finke J, Peschel C, Duyster J, Poeck H, Zeiser R, von Bubnoff N. Activity of therapeutic JAK 1/2 blockade in graft-versus-host disease. Blood. 2014 Jun 12;123(24):3832-42. doi: 10.1182/blood-2013-12-543736. Epub 2014 Apr 7. PMID 24711661
- [Background] Ferrara JL, Levine JE, Reddy P, Holler E. Graft-versus-host disease. Lancet. 2009 May 2;373(9674):1550-61. doi: 10.1016/S0140-6736(09)60237-3. Epub 2009 Mar 11. PMID 19282026
- [Background] Blazar BR, Murphy WJ, Abedi M. Advances in graft-versus-host disease biology and therapy. Nat Rev Immunol. 2012 May 11;12(6):443-58. doi: 10.1038/nri3212. PMID 22576252
- [Result] Kim SH, Ahn J, Ock M, Shin S, Park J, Luo N, Jo MW. The EQ-5D-5L valuation study in Korea. Qual Life Res. 2016 Jul;25(7):1845-52. doi: 10.1007/s11136-015-1205-2. Epub 2016 Mar 10. PMID 26961008
- [Result] Lee SJ, Wolff D, Kitko C, Koreth J, Inamoto Y, Jagasia M, Pidala J, Olivieri A, Martin PJ, Przepiorka D, Pusic I, Dignan F, Mitchell SA, Lawitschka A, Jacobsohn D, Hall AM, Flowers ME, Schultz KR, Vogelsang G, Pavletic S. Measuring therapeutic response in chronic graft-versus-host disease. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: IV. The 2014 Response Criteria Working Group report. Biol Blood Marrow Transplant. 2015 Jun;21(6):984-99. doi: 10.1016/j.bbmt.2015.02.025. Epub 2015 Mar 19. PMID 25796139
- [Result] Zeiser R, Polverelli N, Ram R, Hashmi SK, Chakraverty R, Middeke JM, Musso M, Giebel S, Uzay A, Langmuir P, Hollaender N, Gowda M, Stefanelli T, Lee SJ, Teshima T, Locatelli F; REACH3 Investigators. Ruxolitinib for Glucocorticoid-Refractory Chronic Graft-versus-Host Disease. N Engl J Med. 2021 Jul 15;385(3):228-238. doi: 10.1056/NEJMoa2033122. PMID 34260836
- [Result] Miklos DB, Abu Zaid M, Cooney JP, Albring JC, Flowers M, Skarbnik AP, Yakoub-Agha I, Ko BS, Bruno B, Waller EK, Yared J, Sohn SK, Bulabois CE, Teshima T, Jacobsohn D, Greinix H, Mokatrin A, Lee Y, Wahlstrom JT, Styles L, Socie G. Ibrutinib for First-Line Treatment of Chronic Graft-Versus-Host Disease: Results From the Randomized Phase III iNTEGRATE Study. J Clin Oncol. 2023 Apr 1;41(10):1876-1887. doi: 10.1200/JCO.22.00509. Epub 2023 Jan 6. PMID 36608310
- See also: Pharmaceutical Safety Korea, Jakavi Tablets (Ruxolitinib Phosphate) Precautions for Use and Approved Dosage and Administration (Accessed Oct 19, 2023) — https://nedrug.mfds.go.kr/pbp/CCBBB01/getItemDetailCache?cacheSeq=201301665aupdateTs2023-07-04%2014:51:32.553738b
- See also: ECOG-ACRIN, ECOG Performance Status Scale, Accessed Oct 19 2023 — https://ecog-acrin.org/resources/ecog-performance-status
- See also: National Center for Biotechnology Information (nih,gov), Glucocorticoid Equivalencies, Accessed Oct 19 2023 — https://www.ncbi.nlm.nih.gov/books/NBK279156/table/adrenal_glucocorticoid-therapy-and-adrenal-suppression.T./